CLINICAL TRIAL: NCT05054413
Title: Key Elements for Standardized Reporting in Prostate Cancer Management: An Expert Delphi Consensus Study
Brief Title: Formulating Expert Consensus Guidelines in Cancer Care Using the Delphi Method
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1096; NCI-2021-01928 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1096 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-03-21; First posted 2021-09-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaire): Participants complete 3-4 rounds of questionnaires over 20-30 minutes each over 2 weeks.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study formulates consensus agreement on clinical key elements related to prostate cancer care that are critical for standardization and global reported using a robust Delphi technique, completely remote and electronic. The goal of this survey study is to have a panel of specialty-specific experts create a consensus agreement on a minimum set of key data elements for use in standardized reports. These recommendations would be used to develop standardized methods to report key data in electronic health records to better manage cancer patients at time of diagnosis, treatment, follow up, and into survivorship.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To formulate consensus agreement on a minimum set of clinical key elements that should be included in standardized reports in electronic health records when managing patients with prostate cancer.

OUTLINE:

Participants complete 3-4 rounds of questionnaires over 20-30 minutes each over 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and above
* Board certification in Radiation Oncology, Radiation Physics, Urology, and/or Medical Oncology
* Maintenance of an active practice that includes prostate cancer patients
* English speaking

Exclusion Criteria:

* Medical providers that are not board certified in the professions and/or those who do not treat prostate cancer
* Prisoners, children, and adults unable to consent to participation will also be excluded
* No exclusions were made based on sex, age, racial/ethnic background, or pregnancy status

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with board certification in Radiation Oncology, Radiation Physics, Urology, and/or Medical Oncology
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
To establish a standardized methods to report key data in electronic health records to better manage cancer patients at time of diagnosis, treatment, follow up, and into survivor-ship. | through study completion, an average of a year.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Moreno, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org